CLINICAL TRIAL: NCT00681395
Title: Study to Compare the Bioavailability of ABT-335 and Rosuvastatin From ABT-143 Relative to That From the Co-administration of ABT-335 and Rosuvastatin Calcium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-360
Record Dates: First submitted 2008-05-19; First posted 2008-05-21 (Estimated); Last update posted 2012-09-28 (Estimated); Status verified 2012-09

CONDITIONS: Adverse Events; Pharmacokinetic
MeSH Terms: interventions — 2-(4-(4-chlorobenzoyl)phenoxy)-2-methylpropanoic acid; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): ABT-143 capsules 20/135 mg
  Interventions: Drug: ABT-143
- 2 (Active Comparator): ABT-335 135mg and rosuvastatin 20mg
  Interventions: Drug: ABT-335; Drug: Rosuvastatin
- 3 (Experimental): ABT-143 capsules 5/45mg
  Interventions: Drug: ABT-143
- 4 (Active Comparator): ABT-335 45mg and rosuvastatin 5mg
  Interventions: Drug: ABT-335; Drug: Rosuvastatin

INTERVENTIONS:
Drug: ABT-143 — once daily for 6 days
  Arms: 1; 3
Drug: ABT-335 — once daily for six days
  Arms: 2; 4
Drug: Rosuvastatin — Once daily for 6 days
  Arms: 2; 4

SUMMARY:
To evaluate safety and compare the pharmacokinetic parameters from the fixed dose combination ABT-143 relative to that from the co-administration of the two monotherapies.

ELIGIBILITY:
Inclusion Criteria:

* General good health
* BMI 19 to 29

Exclusion Criteria:

* Currently enrolled in another study
* Females who are pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2008-05; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Adverse event and safety laboratory assessments | 7 days
Pharmacokinetic parameters | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Torbjörn Lundström, MD, Study Director — AstraZeneca
Locations (1):
- Site Reference ID/Investigator# 8089, Orlando, Florida, United States